CLINICAL TRIAL: NCT04065386
Title: Transcutaneous Auricular Vagal Nerve Stimulation for Post-coma Patients With Disorders of Consciousness: a Randomized Double-blind Controlled Trial
Brief Title: Transcutaneous Auricular Vagal Nerve Stimulation for Post-coma Patients With Disorders of Consciousness
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Aurore Thibaut, PhD, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019/91
Record Dates: First submitted 2019-08-21; First posted 2019-08-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Consciousness Disorder; Minimally Conscious State; Vegetative State
Keywords: Vagus nerve stimulation; Transcutaneous electrical nerve stimulation; Non-invasive brain stimulation; Neuromodulation; High-density EEG; Unresponsive wakefulness syndrome; Vegetative state; Minimally Conscious state; Consciousness disorder
MeSH Terms: conditions — Consciousness Disorders; Persistent Vegetative State

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active taVNS (Active Comparator): Patients will receive 5 days of transcutaneous auricular vagal nerve stimulation (taVNS) bilaterally, at the cymba conchae, the active localization.
  It will be preceded and followed by a clinical assessment (Coma Recovery Scale- Revised) and a neurophysiological assessment (128/256 channels EEG and electrocardiograph) the first and last day of stimulation.
  Interventions: Device: Active taVNS
- Sham taVNS (Placebo Comparator): Patients will receive 5 days of transcutaneous auricular vagal nerve stimulation (taVNS) bilaterally, at the ear lobe, the sham localization.
  It will be preceded and followed by a clinical assessment (Coma Recovery Scale- Revised) and a neurophysiological assessment (128/256 channels EEG and electrocardiograph) the first and last day of stimulation.
  Interventions: Device: sham taVNS

INTERVENTIONS:
Device: Active taVNS — Patients will receive transcutaneous auricular vagal nerve stimulation (taVNS) for 5 consecutive days, at the cymba conchae, bilaterally, during 45 minutes (alternating 30 s on and 30 s off periods). Current intensity: 3 mA or less according to the participant's pain threshold, width: 200-300 μsec.
  Arms: Active taVNS
Device: sham taVNS — Patients will receive transcutaneous auricular vagal nerve stimulation (taVNS) for 5 consecutive days, at the ear lobe, bilaterally, during 45 minutes (alternating 30 s on and 30 s off periods). Current intensity: 3 mA or less according to the participant's pain threshold, width: 200-300 μsec.
  Arms: Sham taVNS

SUMMARY:
Non-invasive brain stimulations techniques have recently shown promising results in patients with disorders of consciousness. Notably, a case reported improvement of level of consciousness using transcutaneous auricular vagal nerve stimulation in a patient in unresponsive wakefulness syndrome.

Here we aim to assess the effects of transcutaneous auricular vagal nerve stimulation on post-coma patients with disorders of consciousness in a first randomized controlled trial. To measure these effects, behavioral (Coma recovery scale revised - CRS-R -primary outcome) and neuro-electrophysiological (electroencephalography - EEG - secondary outcome) data will be recorded in severely brain-injured patients with DOC.

DETAILED DESCRIPTION:
Currently, therapeutic options for severely brain-injured patients with disorders of consciousness (DOC), including patients in unresponsive wakefulness syndrome (UWS) and minimally conscious state (MCS), are limited and still need to be improved to influence long-term outcomes. Non-invasive brain stimulations (NIBS) techniques have recently shown promising results in DOC.

Transcutaneous auricular vagal nerve stimulation (taVNS-R, tVNS Technologies GmbH, Germany) seems to be a promising approach. In a recent case report, a patient in UWS improved to MCS using this therapeutic technique.

To confirm this positive result, we propose a first randomized double-blind controlled trial. The patients will be randomized in the active stimulation group and will receive bilateral stimulations of the cymba conchae or in the sham stimulation group and will receive bilateral stimulations of the ear lobe. All stimulations will be performed for 45 minutes bilaterally for 5 consecutive days, between 7 and 90 days post-injury in severely brain-damaged patients with disorders of consciousness. The stimulation will start at 3 mA and will be decreased if signs of pain were observed (more than 4/9 according to the Nociceptive Coma Scale-Revised - NCS-R) until stimulation stays under pain threshold.

Behavioral assessments will be performed using the Coma Recovery Scale-Revised before and after the first and last session by an investigator blinded to the treatment allocation. Fifteen minutes of high-density EEG will also be recorded directly before and after the first and last stimulation session. During this same period of time, electrocardiography (EKG) will be recorded to measure parasympathetic indirect signs of vagal stimulation.

3 months after the last stimulation session, an outcome follow-up will be done, using the Glasgow Outcome Scale Extended (GOS-E) and the Disability Rating scale (DRS).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* State of consciousness: unresponsive wakefulness syndrome (UWS) and minimally conscious state (MCS) as defined by CRS-R performed during the screening period.
* Cerebral damage of known etiology
* Time since injury between 7 and 90 days
* Intact skin at the ears
* Consent given by the substitute decision maker

Exclusion Criteria:

* Anyone who is deemed medically unsuitable for this study as determined by a physician involved with the study (e.g. severe rythmic heart condition)
* Previous history of neurological disorders
* Documented pregnancy
* Active implant (i.e. pacemaker)
* Profound sedation such as one caused by general anaesthetics (e.g., propofol) or a combination of central acting sedatives (e.g., benzodiazepines, opioids)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-02-09 (Actual); Primary Completion 2024-09-21 (Actual); Study Completion 2024-12-21 (Estimated)

PRIMARY OUTCOMES:
Change in CRS-R total score and index score | Before the installation of the EEG equipment in the pre-stimulation period and 5 minutes after the post-stimulation resting state EEG (immediately after removing the equipment).
  Behavioral improvement measured by standardized scale. This scale is ranging from 0 to 23, highest score represents more signs of consciousness. The index score is ranging from 0 to 100.

SECONDARY OUTCOMES:
Change in EEG | 15 min before the stimulation period and 15 min after the stimulation period.
  Improvement in cerebral activity (i.e. power spectrum in the alpha and theta band and connectivity) as measured by EEG

CONTACTS AND LOCATIONS:
Overall Officials: Aurore Thibaut, PhD, Principal Investigator — Université de Liège
Locations (2):
- Belgium (2):
  - Centre Neurologique William Lennox, Ottignies-Louvain-la-Neuve, Brabant Wallon
  - Centre Hospitalier Universitaire de Liège, Liège

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yu YT, Yang Y, Wang LB, Fang JL, Chen YY, He JH, Rong PJ. Transcutaneous auricular vagus nerve stimulation in disorders of consciousness monitored by fMRI: The first case report. Brain Stimul. 2017 Mar-Apr;10(2):328-330. doi: 10.1016/j.brs.2016.12.004. Epub 2016 Dec 14. No abstract available. PMID 28017322
- [Background] Yakunina N, Kim SS, Nam EC. Optimization of Transcutaneous Vagus Nerve Stimulation Using Functional MRI. Neuromodulation. 2017 Apr;20(3):290-300. doi: 10.1111/ner.12541. Epub 2016 Nov 29. PMID 27898202
- [Derived] Vitello MM, Briand MM, Ledoux D, Annen J, El Tahry R, Laureys S, Martin D, Gosseries O, Thibaut A. Transcutaneous vagal nerve stimulation to treat disorders of consciousness: Protocol for a double-blind randomized controlled trial. Int J Clin Health Psychol. 2023 Apr-Jun;23(2):100360. doi: 10.1016/j.ijchp.2022.100360. Epub 2022 Nov 29. PMID 36467262